CLINICAL TRIAL: NCT03458923
Title: Intravitreal Diclofenac Versus Intravitreal Ranibizumab for the Treatment of Diabetic Macular Edema.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Iyad Adnan Salem Goussous, Doctor Iyad Adnan Salem Goussous, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Iyad Goussous
Record Dates: First submitted 2018-02-26; First posted 2018-03-08 (Actual); Last update posted 2018-03-08 (Actual); Status verified 2018-03

CONDITIONS: Diabetic Macular Edema
Keywords: Diclofenac; Ranibizumab; Diabetic Macular Edema
MeSH Terms: interventions — Diclofenac; Anti-Inflammatory Agents, Non-Steroidal; Ranibizumab; Solutions; Injections

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (Active Comparator): 15 eyes will receive 0.1 ml containing 500µg of diclofenac intravitreally, repeated monthly for 3 months.
  Interventions: Drug: Diclofenac Sodium 0.1 ml containing 500µg
- Group B (Active Comparator): 15 eyes will receive 0.5 mg Ranibizumab intravitreally, repeated monthly for 3 months.
  Interventions: Drug: Ranibizumab 0.5 mg Solution for Injection

INTERVENTIONS:
Drug: Diclofenac Sodium 0.1 ml containing 500µg — 15 eyes will receive intravitreal 0.1 ml containing 500µg of Diclofenac Sodium monthly for three months
  Other Names: nonsteroidal anti-inflammatory drug
  Arms: Group A
Drug: Ranibizumab 0.5 mg Solution for Injection — 15 eyes will receive intravitreal 0.5 mg of Ranibizumab monthly for three months
  Other Names: anti vascular endothelial growth factor
  Arms: Group B

SUMMARY:
The study aims to compare the effect of intravitreal non steroidal anti inflammatory (Diclofenac) versus the standard treatment of diabetic macular edema, intravitreal anti vascular endothelial growth factor (Ranibizumab), measuring central macular thickness changes and best corrected visual acuity.

DETAILED DESCRIPTION:
Thirty eyes of diabetic patients with diabetic retinopathy with macular edema will be randomized using simple randomization method into two groups; A and B.

Group A will undergo intravitreal injection of 500µg Diclofenac, repeated monthly for 3 months. Electroretinogram will be performed before the injections, 4 weeks after first injection and 4 weeks after third injection to assess any risk of toxicity.

Colored photography and fundus fluorescein angiography will be done before the first injection to assess the extent of macular leakage at late phases, and to exclude cases with macular ischemia.

Optical coherence tomography will be done to measure the central macular thickness, before the first injection, and before each injection.

Visual acuity will be assessed before and after each injection.

Group B will undergo intravitreal injection of 0.5 mg Ranibizumab, repeated monthly for 3 months. Colored photography and fundus fluorescein angiography will be done before the first injection to assess the extent of macular leakage at late phases, and to exclude cases with macular ischemia.

Optical coherence tomography will be done to measure the central macular thickness, before the first injection, and before each injection.

Visual acuity will be assessed before and after each injection.

All patients will be examined weekly for one month and then monthly for three months after the injection. At every visit, visual acuity, intraocular pressure, and a dilated fundus examination will be performed.

All patients will be required to instill topical antibiotic Gatifloxacin postoperatively 3 times per day for 5 days.

Patients will be warned about the signs and symptoms of complications (endophthalmitis, retinal detachment, vitreous hemorrhage, lens trauma) and asked to seek medical attention immediately.

ELIGIBILITY:
Inclusion Criteria:

1. Diabetic retinopathy with non tractional maculopathy, where central macular thickness is greater than 400µm, with and without cystic changes.
2. Diabetes Mellitus type one and two
3. Best Corrected Visual Acuity > 0.1 LogMar

Exclusion Criteria:

1. Patients treated with diclofenac, Ranibizumab or Bevacizumab in the past 3 months
2. Patients with a history of branch or central retinal artery occlusion
3. Patients without clear media and adequate pupillary dilation that allows proper fundoscopy and imaging, and patients who are not complaint with the regular visits.
4. Visual Significant Cataract
5. Evidence of vitreomacular traction or macular ischemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-01 (Actual); Primary Completion 2018-06 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Change in best corrected visual acuity | 3 months of follow up
  Measuring the best corrected visual acuity
Change in central macular thickness | 3 months of follow up
  Measuring the change in central macular thickness using Optical Coherence Tomography

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed S El Agha, PhD, Study Chair — Cairo University
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided